CLINICAL TRIAL: NCT01591551
Title: NAPS-MS: NAtalizumab Effects on Parameters of Sleep in Patients With Relapsing Forms of Multiple Sclerosis Experiencing Fatigue or Sleepiness
Brief Title: NAPS-MS: NAtalizumab Effects on Parameters of Sleep in Patients With Multiple Sclerosis Experiencing Fatigue or Sleepiness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cornerstone Health Care, PA (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: US-TYS-11-10221
Record Dates: First submitted 2012-04-22; First posted 2012-05-04 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab (Tysabri) naive (Other): Patients who are newly prescribed Natalizumab (TYSABRI®), but have not received their first infusion, will be invited to participate.
  Interventions: Drug: Natalizumab (Tysabri)

INTERVENTIONS:
Drug: Natalizumab (Tysabri) — 300 mg IV every 4 weeks

SUMMARY:
The purpose of this study is to assess the impact of Natalizumab (Tysabri) therapy on sleep efficiency, total sleep time and sleep latency, in Multiple Sclerosis (MS) patients receiving Natalizumab for 6 months relative to baseline.

DETAILED DESCRIPTION:
Natalizumab has been shown to positively impact fatigue and cognition. The mechanism by which this occurs is unknown. Change in quality of sleep is one possible etiology of these findings. This study will help to elucidate the mechanisms that lead to reduced fatigue/sleepiness and less cognitive dysfunction in MS patients who go on Natalizumab therapy. Understanding these factors may help neurologists better differentiate between the different therapeutic options for MS and how they may impact symptoms that negatively affect quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing form of multiple sclerosis
* Able to give informed consent and committed to follow the protocol
* EDSS from 0 to 6.0
* Epworth Sleepiness Scale > 9 or Modified Fatigue Impact Scale > 30 or Fatigue Severity Scale > 4
* Age range of 18 - 65 years of age
* Naïve to Natalizumab
* Enrolled in the TOUCH program

Exclusion Criteria:

* Severe cognitive impairment
* Coexisting severe medical condition
* Inability to speak English or read
* Inability to give valid informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in parameters of sleep as measured by polysomnography and multi-sleep latency test over 6 months of Natalizumab treatment. | Baseline and 6 months

SECONDARY OUTCOMES:
Change in neurocognition parameters over 6 months of Natalizumab treatment and correlation with changes in sleep efficiency. | Baseline and 6 months
Change in subjective measures of fatigue, sleepiness and mood over 6 months of Natalizumab treatment and correlation with changes in sleep efficiency. | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Sater, MD, PhD, Principal Investigator — Cornerstone Healthcare
Locations (3):
- United States (3):
  - South Shore Neurologic Associates, Patchogue, New York
  - Cornerstone Neurology, High Point, North Carolina
  - Providence Brain Institute, Portland, Oregon